CLINICAL TRIAL: NCT07001111
Title: Investigation of the Effectiveness of Kinesiological Taping in Cubital Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Feyza Nur Yucel, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-17
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cubital Tunnel Syndrome; Kinesio Taping; Ulnar Neuropathies
Keywords: Cubital Tunnel Syndrome; Kinesio taping; ulnar neuropathies
MeSH Terms: conditions — Cubital Tunnel Syndrome; Ulnar Neuropathies | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Prospective Experimental (Randomized Controlled) Study
Who Masked: Participant
Masking Description: The study is designed as a single-blind trial, where patients will be blinded to the treatment group they are assigned to. In order to assess the effectiveness of the treatment, it is essential that the patient is unaware of being in the placebo group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): All patients will be provided with information and an exercise sheet containing pictures on ulnar nerve gliding exercises. To monitor whether patients are performing the exercises correctly, they will be asked to come to the hospital once a week, where they will perform the exercises under the supervision of a physiotherapist. In the exercise program, different positions will be held for 30 seconds, with a 1-minute rest between them, and the exercises will be performed twice a day .
  Interventions: Other: Ulnar nerve mobilization exercise; Diagnostic Test: Numeric Rating Scale (NRS); Diagnostic Test: the ulnar nerve cross-sectional area measured by ultrasound; Diagnostic Test: Neuropathic pain scale (measured using the DN-4 scale); Diagnostic Test: SF-12 Quality of Life Scale; Diagnostic Test: QUICK-DASH; Diagnostic Test: Grip strength measured with a hand dynamometer
- Kinesio Taping (Active Comparator): It will be applied once a week for 3 weeks to the affected elbow by an experienced practitioner. During taping, the space correction technique will be used. In this technique, the kinesiological tape is applied with a hole cut in the center, slightly larger than the area to be treated .
  Interventions: Other: kinesio taping; Other: Ulnar nerve mobilization exercise; Diagnostic Test: Numeric Rating Scale (NRS); Diagnostic Test: the ulnar nerve cross-sectional area measured by ultrasound; Diagnostic Test: Neuropathic pain scale (measured using the DN-4 scale); Diagnostic Test: SF-12 Quality of Life Scale; Diagnostic Test: QUICK-DASH; Diagnostic Test: Grip strength measured with a hand dynamometer
- Sham Taping (Sham Comparator): It will be applied in the same way as kinesiological taping with adhesive tape.
  Interventions: Other: Ulnar nerve mobilization exercise; Other: Sham (No Treatment); Diagnostic Test: Numeric Rating Scale (NRS); Diagnostic Test: the ulnar nerve cross-sectional area measured by ultrasound; Diagnostic Test: Neuropathic pain scale (measured using the DN-4 scale); Diagnostic Test: SF-12 Quality of Life Scale; Diagnostic Test: QUICK-DASH; Diagnostic Test: Grip strength measured with a hand dynamometer

INTERVENTIONS:
Other: kinesio taping — Kinesio taping at the level of the cubital tunnel on the elbow
  Arms: Kinesio Taping
Other: Ulnar nerve mobilization exercise — All patients will be provided with information and an exercise sheet containing pictures on ulnar nerve gliding exercises. To monitor whether patients are performing the exercises correctly, they will be asked to come to the hospital once a week, where they will perform the exercises under the supervision of a physiotherapist. In the exercise program, different positions will be held for 30 seconds, with a 1-minute rest between them, and the exercises will be performed twice a day .
Other: Sham (No Treatment) — It will be applied in the same way as kinesiological taping with adhesive tape.
  Arms: Sham Taping
Diagnostic Test: Numeric Rating Scale (NRS) — Description: To demonstrate that kinesiological taping will result in a reduction of pain intensity associated with Cubital Tunnel Syndrome, as measured by the Numeric Rating Scale (NRS) ranging from 0 to 10.
Diagnostic Test: the ulnar nerve cross-sectional area measured by ultrasound — The measurements will be taken with the patient in a supine position, the affected arm in shoulder abduction and external rotation, and the elbow flexed at 70°-90°. After applying a generous amount of gel, the lateral edge of the ultrasound probe will be placed on the medial epicondyle, and the medial edge of the probe will be positioned on the olecranon; the ulnar nerve will be directly examined in the retroepicondylar groove. Once the nerve is visualized, the widest point will be identified, and cross-sectional area (CSA) measurements will be taken with the probe perpendicular to the nerve at the center of the screen . The measurements will be repeated twice, and the average will be calculated.
Diagnostic Test: Neuropathic pain scale (measured using the DN-4 scale) — The DN4 questionnaire consists of two main sections and a total of ten questions. The first section includes seven questions related to pain characteristics and sensory information obtained through patient interview. These questions are about burning, electric shocks, coldness, tingling, pricking, numbness, and itching. The second section contains three statements related to physical examination (touch hypoesthesia, pinprick hypoesthesia, and allodynia). For each statement, "yes" or "no" responses are given. A score of "1" is assigned for "yes" answers and "0" for "no" answers, and the scores are summed. A total score of 4 or more out of 12 is interpreted as neuropathic pain.
Diagnostic Test: SF-12 Quality of Life Scale — The SF-12 Quality of Life Scale is a short form of the SF-36 Quality of Life Scale. While the SF-36 is used for chronic conditions (states), the SF-12 is used for short-term assessments (clinical findings). Similarly, it is also used to gather information about the patient's general health status. The SF-12 provides the same summary component scores as the SF-36, but with fewer items, making it a significant advantage due to its shorter application time. The scale asks the patient about their health opinions, how they feel, and how easily they can perform their usual activities. Scores range from 0 to 100, with higher scores indicating better quality of life.
Diagnostic Test: QUICK-DASH — QUICK-DASH (Shoulder, Arm, and Hand Problems Questionnaire):
  This questionnaire assesses both the ability to perform certain physical activities as well as the symptoms of the disease. Each question is answered based on the condition of the past week, and the appropriate score is marked. The answer is given based solely on the ability to perform the physical activity, without considering which hand or arm is injured.
  Scoring:
  1. = No difficulty
  2. = Mild difficulty
  3. = Moderate difficulty
  4. = Severe difficulty
  5. = Unable to perform
  QUICK DASH DISABILITY/SYMPTOM SCORE:
  ([(n total score] - 1) x 25; where n represents the number of questions answered. If more than one question is unanswered, the Quick DASH score cannot be calculated.
  SCORE FOR OPTIONAL MODELS:
  For each model, divide the total score by 4, subtract 1, and multiply by 25. If more than one question is unanswered, the score for optional models cannot be calculated.
  Based on the results of the questionnaire, a score b
Diagnostic Test: Grip strength measured with a hand dynamometer — Grip strength will be measured using a hand dynamometer, with the average of three measurements taken, each followed by a 30-second rest period.

SUMMARY:
This study aims to investigate the effect of kinesiological taping, applied in addition to exercise, on clinical symptoms in patients diagnosed with Cubital Tunnel Syndrome. The patients will be randomized into three groups (exercise, exercise + kinesiological taping, exercise + sham taping) and will be evaluated at the 1st and 3rd months after a 3-week treatment period.

DETAILED DESCRIPTION:
Cubital Tunnel Syndrome (CuTS), characterized by the compression of the ulnar nerve at the elbow, is a condition that causes symptoms such as pain, numbness, paresthesia, and muscle weakness in the affected limb. Ulnar nerve compression is the second most common entrapment neuropathy after median nerve entrapment . The ulnar nerve can become compressed at various locations, including the elbow and wrist. The nerve is formed by the C8 and T1 spinal nerve roots, which make up the lower trunk and medial cord of the brachial plexus. It travels along the medial aspect of the humerus, passes through Struthers' arcade, the retro-epicondylar groove, and enters the cubital tunnel. The roof of the cubital tunnel is known as the cubital tunnel retinaculum. The ulnar nerve then passes beneath the aponeurosis of the flexor carpi ulnaris muscle and its two heads, where the upper edge of the aponeurosis forms the Osborne ligament, which is likely the most commonly affected area in ulnar nerve entrapment. In the forearm, the ulnar nerve is located beneath the flexor carpi ulnaris muscle and innervates this muscle along with the ulnar half of the flexor digitorum profundus muscle. The nerve then proceeds toward Guyon's canal along with the ulnar artery. Distally, the nerve branches into three divisions: the dorsal sensory branch, the volar superficial sensory branch, and the deep motor branch. The deep motor branch descends into the deep part of the hand beneath the edge of the aponeurosis surrounding the hook of the hamate bone, innervating most of the hypothenar and intrinsic muscles. The dorsal sensory branch leaves the main trunk approximately 5-8 cm proximal to Guyon's canal and innervates the dorsal ulnar portion of the hand .

In patients with Cubital Tunnel Syndrome, pain, numbness, paresthesia in the 4th and 5th fingers, and in advanced stages, muscle weakness leading to atrophy of the hypothenar muscles and claw hand deformity may be observed. The diagnosis is made through electrophysiological studies (EMG/NCS).

Treatment options include both conservative and surgical approaches. Surgical options include cubital tunnel decompression, medial epicondylectomy, and ulnar nerve transposition . Surgical treatment is generally preferred for patients with muscle weakness and atrophy, as well as those who do not respond to conservative treatments. Conservative treatment options include avoiding positions of the elbow that may exacerbate symptoms, splinting, exercise, electrotherapy, and local steroid injections .

Kinesiotaping, developed by chiropractor and acupuncturist Kenzo Kase in the late 1970s, is a commonly used conservative treatment option for musculoskeletal pathologies in physical therapy clinics. The tape is made of cotton, stretches longitudinally up to 40%, is water-resistant, and can stay on the skin for up to 7 days.

Kinesiotaping is believed to support muscles, correct joint movement, enhance blood and lymph circulation, provide proprioceptive input, and reduce pain and muscle spasms . Various physical therapy modalities, steroid injections, and dry needling have been studied for their effects on Cubital Tunnel Syndrome. Kinesiotaping has been shown to be effective in patients with Carpal Tunnel Syndrome. However, there is no study available on the use of kinesiotaping in CuTS patients. This simple, cost-effective treatment modality, commonly used in physical therapy practice for various pathologies, will be investigated for its efficacy in patients with Cubital Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Patients with at least 3 points of pain according to the Numeric Rating Scale (NRS)
* Patients diagnosed with Cubital Tunnel Syndrome via Electroneuromyography (ENMG)
* Literate
* Willing to consent to participate in the study

Exclusion Criteria:

* Having any secondary entrapment neuropathy such as diabetes, inflammatory arthritis, or hypothyroidism
* Pregnancy
* Active cancer presence
* Skin infection, burns, wounds, or scars on the forearm
* History of elbow trauma
* Cervical radiculopathy or brachial plexopathy
* Polyneuropathy
* Having previously undergone Cubital Tunnel decompression surgery
* Having received a corticosteroid injection into the Cubital Tunnel within the last 3 months
* Illiterate
* Not consenting to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 3 months
  To demonstrate that kinesiological taping will result in a reduction of pain intensity associated with Cubital Tunnel Syndrome, as measured by the Numeric Rating Scale (NRS) ranging from 0 to 10.

SECONDARY OUTCOMES:
the ulnar nerve cross-sectional area measured by ultrasound | 3 months
  The measurements will be taken with the patient in a supine position, the affected arm in shoulder abduction and external rotation, and the elbow flexed at 70°-90°. After applying a generous amount of gel, the lateral edge of the ultrasound probe will be placed on the medial epicondyle, and the medial edge of the probe will be positioned on the olecranon; the ulnar nerve will be directly examined in the retroepicondylar groove. Once the nerve is visualized, the widest point will be identified, and cross-sectional area (CSA) measurements will be taken with the probe perpendicular to the nerve at the center of the screen .
  The measurements will be repeated twice, and the average will be calculated.
Neuropathic pain scale (measured using the DN-4 scale | 3 months
  The DN4 questionnaire consists of two main sections and a total of ten questions. The first section includes seven questions related to pain characteristics and sensory information obtained through patient interview. These questions are about burning, electric shocks, coldness, tingling, pricking, numbness, and itching. The second section contains three statements related to physical examination (touch hypoesthesia, pinprick hypoesthesia, and allodynia). For each statement, "yes" or "no" responses are given. A score of "1" is assigned for "yes" answers and "0" for "no" answers, and the scores are summed. A total score of 4 or more out of 12 is interpreted as neuropathic pain.
SF-12 Quality of Life Scale | 3 months
  The SF-12 Quality of Life Scale is a short form of the SF-36 Quality of Life Scale. While the SF-36 is used for chronic conditions (states), the SF-12 is used for short-term assessments (clinical findings). Similarly, it is also used to gather information about the patient's general health status. The SF-12 provides the same summary component scores as the SF-36, but with fewer items, making it a significant advantage due to its shorter application time. The scale asks the patient about their health opinions, how they feel, and how easily they can perform their usual activities. Scores range from 0 to 100, with higher scores indicating better quality of life.
QUICK-DASH | 3 months
  QUICK-DASH (Shoulder, Arm, and Hand Problems Questionnaire):
  This questionnaire assesses both the ability to perform certain physical activities as well as the symptoms of the disease. Each question is answered based on the condition of the past week, and the appropriate score is marked. The answer is given based solely on the ability to perform the physical activity, without considering which hand or arm is injured.
  Scoring:
  1. = No difficulty
  2. = Mild difficulty
  3. = Moderate difficulty
  4. = Severe difficulty
  5. = Unable to perform
  QUICK DASH DISABILITY/SYMPTOM SCORE:
  ([(n total score] - 1) x 25; where n represents the number of questions answered. If more than one question is unanswered, the Quick DASH score cannot be calculated.
  SCORE FOR OPTIONAL MODELS:
  For each model, divide the total score by 4, subtract 1, and multiply by 25. If more than one question is unanswered, the score for optional models cannot be calculated.
  Based on the results of the questionnaire, a score b
Grip strength measured with a hand dynamometer | 3 months
  Grip strength will be measured using a hand dynamometer, with the average of three measurements taken, each followed by a 30-second rest period.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Health Sciences University, Istanbul, Uskudar
  - Sultan 2. Abdülhamid Han Eğitim ve Araştırma Hastanesi, Istanbul, Üsküdar

IPD SHARING:
Plan to Share IPD: No
Data sharing not planned

REFERENCES:
- [Background] Stewart JD. The variable clinical manifestations of ulnar neuropathies at the elbow. J Neurol Neurosurg Psychiatry. 1987 Mar;50(3):252-8. doi: 10.1136/jnnp.50.3.252. PMID 3031220